CLINICAL TRIAL: NCT07311850
Title: Evaluating The Efficacy and Safety of MET097, a Fully-Biased, Ultra Long-Acting GLP-1RA, In People With Overweight or Obesity: A Phase 3, Multi-Center Randomized, Controlled Trial (VESPER-4)
Brief Title: Efficacy and Safety of MET097 Once-Weekly in People With Overweight or Obesity
Acronym: VESPER-4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Metsera, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MET097-25-301
Record Dates: First submitted 2025-12-29; First posted 2025-12-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MET097 Dose 1 (Experimental): Participants will receive MET097 administered subcutaneously
  Interventions: Drug: MET097
- MET097 Dose 2 (Experimental): Participants will receive MET097 administered subcutaneously
  Interventions: Drug: MET097
- MET097 Dose 3 (Experimental): Participants will receive MET097 administered subcutaneously
  Interventions: Drug: MET097
- Placebo (Placebo Comparator): Once-weekly placebo administered via subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MET097 — Once-weekly MET097 administered via subcutaneous injection
  Other Names: PF-08653944
  Arms: MET097 Dose 1; MET097 Dose 2; MET097 Dose 3
Drug: Placebo — Once-weekly placebo administered via subcutaneous injection
  Arms: Placebo

SUMMARY:
This study investigates the efficacy and safety of once weekly injectable MET097 in adult participants with obesity or overweight with weight-related comorbidities excluding T2D. This trial will last for a duration of 84 weeks. The primary endpoint will be assessed after 64 weeks of treatment with the secondary at 84 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2 or BMI ≥ 27.0 kg/m2 to <30.0 kg/m2 and presence of at least 1 of the following weight- related comorbidities: Hypertension, dyslipidemia, obstructive sleep apnea, or cardiovascular disease)

Exclusion Criteria:

* Have any form of diabetes
* Have a self-reported body weight change > 5 kg (11 pounds) within 3 months prior to Screening
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of chronic pancreatitis or presence of acute pancreatitis within the past 180 days prior to the Screening visit; or active/current, symptomatic gallbladder disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in body weight | Baseline (Day 0) to Week 64

SECONDARY OUTCOMES:
Percentage of Participants who achieve ≥5% of reduction from baseline body weight | Baseline (Day 0) to Week 64
Percentage of Participants who achieve ≥10% of reduction from baseline body weight | Baseline (Day 0) to Week 64
Percentage of Participants who achieve ≥15% of reduction from baseline body weight | Baseline (Day 0) to Week 64
Percentage of Participants who achieve ≥20% of reduction from baseline body weight | Baseline (Day 0) to Week 64
Change from baseline in Fasting triglycerides | Baseline (Day 0) to Week 64
Change from baseline in non-high-density lipoprotein-cholesterol (non-HDL-C) (mg/dL) | Baseline (Day 0) to Week 64
Change from baseline in systolic blood pressure (mmHg) | Baseline (Day 0) to Week 64
Change from baseline in the Short Form 36 health survey (SF-36) physical function domain score | Baseline (Day 0) to Week 64
Mean change from baseline in body weight | Baseline (Day 0) to Week 84

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Research Site 97301-001007, Riverside, California
  - Research Site 97301-001070, Torrance, California
  - Research Site 97301-001077, Englewood, Colorado
  - Research Site 97302-001001, Hollywood, Florida
  - Research Site 97301-001309, Cary, North Carolina